CLINICAL TRIAL: NCT03971318
Title: A Prospective Multicenter Cohort Study on the Efficacy and Safety of Stratified Treatment of Chinese Children With Lymphoblastic Lymphoma Based on Risk Factors
Brief Title: A Prospective Multicenters Clinical Cohort Study of Stratified Treatment of Chinese Children With LBL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiao-Fei Sun, professor, Sun Yat-sen University
Other Study IDs: SCCCG-LBL-2017-001
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Lymphoma, Non-Hodgkin; Lymphoblastic Lymphoma, Childhood; PTEN Loss; NOTCH1 Gene Mutation; Pediatric Cancer
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With the development of molecular biology and precise medical treatment, new challenges have been raised in the diagnosis and treatment of non-Hodgkin lymphoma (NHL) in children. In recent years, the criteria for clinical staging and efficacy evaluation of NHL in children have been updated. Recent clinical studies of COG in the United States and LMB in France have confirmed that molecular biological markers such as Notch1, PTEN and LOH6q are significantly associated with the prognosis of T-lymphoblastic lymphoma (T-LBL). These molecular biological markers should be included in the new risk stratification system. High-intensity treatment of high-risk patients will improve survival. Recent studies have also suggested that PET/CT is helpful in evaluating residual lesions in patients with lymphoma after chemotherapy. In order to keep pace with the times in the diagnosis, clinical staging, risk stratification, efficacy evaluation and treatment of NHL in children. SCCCG-LBL-2017 was formulated by South China Children's Cancer Group of Non-Hodgkin lymphoma, which mainly updated in clinical staging, efficacy evaluation, risk stratification, treatment,etc..

DETAILED DESCRIPTION:
Research purpose:

1. To investigate the efficacy and safety of SCCCG-LBL-2017 in Chinese children with LBL.
2. To explore the feasibility of risk stratification of T-LBL by combining genotyping.
3. To investigate the correlation between MDD and MRD in lymphoblastic lymphoma and prognosis.
4. To investigate the role of PET/CT in the assessment of residual lymphoblastic lymphoma.
5. To explore the effect of reducing HD-MTX dosage and shortening maintenance therapy time on the efficacy and survival of low-risk LBL patients.
6. To explore the effect of prolonging the duration of maintenance therapy on the efficacy and survival of high-risk LBL patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age < 18 years old
2. Pathologically confirmed lymphoblastic lymphoma
3. Newly diagnosed patients
4. Informed consent of guardian of children patients -

Exclusion Criteria:

1. Age > 18 years old
2. Recurrent lymphoblastic lymphoma
3. Secondary immunodeficiency.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: lymphoblastic lymphoma patients#age at diagnosis < 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-05-05 (Actual); Primary Completion 2022-05-05 (Estimated); Study Completion 2025-05-05 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | through study completion, maximal eight years
  EFS is defined as time from start of treatment/randomization up to event or to date of last contact for patients without event. The following occurrences are defined as an event: non-response, progressive disease or relapse, treatment related death, death of any other cause or diagnosis of secondary malignancies.

SECONDARY OUTCOMES:
Overall survival (OS) | through study completion, maximal eight years
  OS is defined as time from start of treatment/randomization up to death of any
Relapse-free survival (RFS) | through study completion, maximal eight years
  RFS is defined as time from start of treatment/randomization up to event or to date of last contact for patients without event. The following occurrences are defined as an event: non-response, progressive disease, or relapse.
Response rate (RR) | on an average 3 weeks after finish of treatment
  Complete response, partial remission, objective effect, stable disease or progressive disease
Adverse event rate | through study completion, maximal eight years
  Rate of patients with acute toxicity defined as grade III/IV/V AE

CONTACTS AND LOCATIONS:
Overall Officials: Zhen zijun, Study Director — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonn BR, Rohde M, Zimmermann M, Krieger D, Oschlies I, Niggli F, Wrobel G, Attarbaschi A, Escherich G, Klapper W, Reiter A, Burkhardt B. Incidence and prognostic relevance of genetic variations in T-cell lymphoblastic lymphoma in childhood and adolescence. Blood. 2013 Apr 18;121(16):3153-60. doi: 10.1182/blood-2012-12-474148. Epub 2013 Feb 8. PMID 23396305
- [Result] Callens C, Baleydier F, Lengline E, Ben Abdelali R, Petit A, Villarese P, Cieslak A, Minard-Colin V, Rullier A, Moreau A, Baruchel A, Schmitt C, Asnafi V, Bertrand Y, Macintyre E. Clinical impact of NOTCH1 and/or FBXW7 mutations, FLASH deletion, and TCR status in pediatric T-cell lymphoblastic lymphoma. J Clin Oncol. 2012 Jun 1;30(16):1966-73. doi: 10.1200/JCO.2011.39.7661. Epub 2012 Apr 30. PMID 22547598